CLINICAL TRIAL: NCT00406809
Title: A Phase 1/2a Study Evaluating the Safety, Pharmacokinetics and Efficacy of ABT-263 in Subjects With Relapsed or Refractory Lymphoid Malignancies
Brief Title: A Study of ABT-263 in Subjects With Relapsed or Refractory Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M06-814; NCT00408811 (obsolete NCT alias)
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Chronic Lymphoid Leukemia; Lymphoid Malignancies; Non-Hodgkin's Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Peripheral T-cell Lymphoma
Keywords: Sezary syndrome; cutaneous T-cell lymphoma; follicular lymphoma; marginal zone lymphoma; indolent T-cell lymphoma; Navitoclax; Non-Hodgkin's lymphoma; peripheral T-cell lymphoma; ABT-263; lymphoid malignancies; chronic lymphoid leukemia; mycosis fungoides; mantle cell lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, T-Cell, Peripheral; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone; Mycosis Fungoides | interventions — navitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1a and 1b (Experimental): Relapsed or refractory lymphoid malignancies
  Interventions: Drug: ABT-263
- Arm A (Phase 2a) (Experimental): Relapsed or refractory follicular lymphoma
  Interventions: Drug: ABT-263
- Arm B (Phase 2a) (Experimental): Relapsed or refractory mantle cell, peripheral T-cell, cutaneous T-cell lymphoma including mycosis fungoides and Sezary syndrome, or other indolent B-cell lymphomas such as marginal zone lymphoma
  Interventions: Drug: ABT-263
- Extension Study (Experimental): Relapsed or refractory follicular lymphoma or Relapsed or refractory mantle cell, peripheral T-cell, cutaneous T-cell lymphoma including mycosis fungoides and Sezary syndrome, or other indolent B-cell lymphomas such as marginal zone lymphoma
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — Oral solution
  Phase 1 dosing was under two different schedules: 14 days on drug, 7 days off or 21 days continuous dosing.
  Oral solution and tablets
  Phase 2a dosing under 21 day continuous dosing.
  - 150 mg lead-in dose for 7-14 days followed by a 325 mg continuous once daily dose.

SUMMARY:
The Phase 1 portion of the study evaluated the pharmacokinetic profile and safety of ABT-263 with the objective of defining the dose limiting toxicity and maximum tolerated dose in subjects with lymphoid malignancies. The Phase 2a portion of the study is evaluating ABT-263 using a step-up dosing regimen and may be increased to the defined recommended Phase 2 dose to obtain additional safety information and a preliminary assessment of efficacy in subject with lymphoid malignancies. The Extension portion of the study is to allow Phase 2a subjects who remain active 1 year after the last subject enrolls or who have been on study approximately 1 year to continue receiving ABT-263 with less frequent study evaluations. Subjects in the Extension Study will continue receiving study drug for up to 7 years after the last subject transitions to the Extension Study, or until disease progression or toxicity that necessitates discontinuation (whichever comes first).

DETAILED DESCRIPTION:
Enrollment breakdown: Entered Study: Phase 1a: 39; Phase 1b: 19; Phase 2a: 33; Total: 91 Entered Treatment: Phase 1a: 38; Phase 1b: 17; Phase 2a: 26; Total: 81

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses:

  * 1a/1b - lymphoid malignancy;
  * 2a, Arm A - follicular lymphoma;
  * 2a, Arm B - mantle cell, peripheral or cutaneous T-cell lymphomas including mycosis fungoides and Sezary syndrome or other indolent B-cell lymphomas such as marginal zone lymphoma;
* Received at least 1 prior chemotherapy treatment regimen (P1a/1b) and relapsed or refractory disease (P2a).
* Eastern Cooperative Oncology Group (ECOG) score of <= 1.
* Magnetic Resonance Imaging (MRI)/computed tomography (CT) negative for subdural or epidural hematoma w/in 28 days prior to first dose, if clinically indicated.
* Stable dose of Selective serotonin reuptake inhibitors (SSRI) antidepressants for at least 21 days prior to 1st dose.
* Adequate bone marrow (BM) independent of any growth factor support (except with heavily infiltrated bone marrow (80% or more)):

  * Absolute Neutrophil Count (ANC) >= 1000/µL;
  * Platelets >= 100,000/mm3 (entry count must be independent of transfusion with in 14 days of Screening);
  * Hemoglobin >= 9.0/dL.
* Adequate coagulation, renal, and hepatic function:

  * Serum creatinine <= 2.0 mg/dL or calculated creatinine clearance >= 50 mL/min;
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 3.0 x Upper Limit of Normal (ULN);
  * Bilirubin <= 1.5 x ULN;
  * Gilbert's Syndrome may have a bilirubin > 1.5 x ULN;
  * Coagulation: Activated partial thromboplastin time (aPTT), Prothrombin Time (PT), not to exceed 1.2 x ULN
* Females must be surgically sterile, postmenopausal (at least 1 year), or negative results for a pregnancy test performed at Screening on a serum sample obtained with in 14 days prior to initial dose, and prior to dosing on a urine sample obtained on C1 D-3 (P1a) or Lead-in D1 (P1b, P2a) if > 7 days since serum results.
* Females not surgically sterile or postmenopausal (at least 1 year) and non-vasectomized males must practice birth control.
* P2a only: History of autologous stem cell transplant must be > 6 months post transplant with adequate BM independent of growth factor support per lab reference range at Screening as follows:

  * Absolute Neutrophil Count (ANC) >= 1,500/µL;
  * Platelets >= 125,000/mm3 (entry platelet count must be independent of transfusion with in 14 days of Screening);
  * Hemoglobin >= 10.0g/dL;
* Measurable disease by International Working Group (IWG)/National Cancer Institute- sponsored Working Group (NCI-WG) criteria.
* At least one of following for Pharmacodynamics (P2a):

  * archived diagnostic Formalin Fixed Paraffin Embedded (FFPE) tumor tissue with no intervening treatment since biopsy,
  * core needle biopsy of malignant lymph node, or
  * bone marrow aspirate or core positive for lymphoma.

Extension Study Inclusion Criteria Phase 2a subjects who enter the Extension Study must continue to meet all Inclusion and Exclusion criteria, with the exception of Inclusion Criterion regarding measurable disease by International Working Group (IWG)/National Cancer Institute- sponsored Working Group (NCI-WG) criteria and Inclusion Criteria regarding laboratory parameters for hematology, coagulation, and chemistry. Subjects entering the Extension Study must also have stable lab values per applicable laboratory reference ranges. In addition, subjects must also meet the following criteria:

* Subjects must meet the following hematology and coagulation lab criteria:

  * Platelet counts must be >= 25,000/mm3 (untransfused). Platelet counts <= 50,000/mm3 must be stable and monitored at an increased frequency at the discretion of the investigator.
  * Absolute Neutrophil count (ANC) >= 500/µL. ANC >= 500/µL and < 1,000/µL should be monitored at an increased frequency at the discretion of the investigator.
  * Hemoglobin of >= 8.0 g/dL.
  * aPTT, PT is not to exceed 1.2 x ULN.
* Chemistry values must not exceed Grade 2. Grade 2 chemistry labs should be monitored at an increased frequency at the discretion of the investigator. Subjects must meet the following chemistry criteria:

  * Serum creatinine <= 3.0 x the upper normal limit (ULN) of institution's normal range. * AST and ALT <= 5.0 x the upper normal limit (ULN) of institution's normal range.
  * Bilirubin <= 3.0 x ULN. Subjects with Gilbert's Syndrome may be allowed to have a Bilirubin > 3.0 x ULN based on a joint decision between the investigator and Abbott medical monitor.

Exclusion Criteria:

* History of, or is, clinically suspicious for cancer-related Central Nervous System (CNS) disease, lymphoid or non-lymphoid.
* Undergone an allogeneic or autologous stem cell transplant.
* Underlying, predisposing condition of bleeding or currently exhibits signs of clinically significant bleeding.
* Recent history of non-chemotherapy induced thrombocytopenic associated bleeding with in 1 year prior to first dose.
* Active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
* Active immune thrombocytopenic purpura or history of being refractory to platelet transfusions with in 1 year prior to first dose.
* Significant history of cardiovascular disease, renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease.
* Females pregnant or breast-feeding.
* Positive for human immunodeficiency virus (HIV)
* History of other active malignancies with in the past 3 years (P1a/1b) or past 5 years (P2a), except adequately treated in situ carcinoma of the cervix uteri; basal or squamous cell carcinoma; in situ carcinoma of the bladder; previous malignancy confined and surgically resected with curative intent.
* Evidence of other clinically significant uncontrolled condition(s), including, but not limited to active systemic fungal infection; diagnosis of fever and neutropenia with in 1 week prior to study drug.
* Received steroid therapy with in 7 days prior to 1st dose of study drug for anti-neoplastic intent.
* Received any anti-cancer therapy, including chemotherapy, immunotherapy, radiotherapy, hormonal or any investigational therapy, with in 14 days prior to first dose of study drug, or has not recovered to <Gr2 clinically significant AE(s) /toxicity(s) of the previous therapy.
* Received a biologic with in 30 days prior to first dose.
* Currently receiving or requires anticoagulation therapy or any drugs or herbal supplements that affect platelet function, with the exception of low-dose anticoagulation medications that are used to maintain the patency of a central venous catheter.
* Received aspirin with in 7 days prior to first dose and during ABT-263 administration.
* Consumed grapefruit or grapefruit products with in 3 days prior to first dose.
* P1a/1b only: Diagnosed with Posttransplant lymphoproliferative disorder (PTLD); Burkitt's, Burkitt-like, or HIV-associate lymphoma; lymphoblastic lymphoma/leukemia; or multiple myeloma.
* Subject has received CYP3A inhibitors (e.g., ketoconazole, clarithromycin) within 7 days prior to the administration of the first dose of ABT-263 (P2a).
* Subject had a prior significant toxicity from another Bcl-2 family protein inhibitor (P2a).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Determine dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended Phase 2 dose (RPTD) and schedule - intermittent dosing. | Repeating sequence of 14 days on therapy and 7 days off.
  1a: Determination of dose limiting toxicity (DLT) and maximum tolerated dose (MTD) under a 14/21 day dosing schedule
Phase 1b: Determine dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended Phase 2 dose (RPTD) and schedule - continuous dosing. | 21 day continuous dosing.
  Phase 1b: Determination of ABT-263 dose limiting toxicity (DLT) and maximum tolerated dose (MTD) under a 21 day continuous dosing schedule.
Phase 2a: Continued assessment of safety profile at the recommended Phase 2 dose (RPTD) and schedule - continuous dosing. | 21 day continuous dosing.
  Phase 2a: Continued assessment of the safety profile of ABT-263 at the Recommended Phase 2 Dose (RPTD) and schedule under a 21 day continuous dosing.
Phase 2a: Assessment of preliminary efficacy signals including biomarker assessment - continuous dosing. | 21 day continuous dosing.
  Phase 2a: Assessment of the preliminary efficacy signals of ABT-263, including biomarker assessment, at the Recommended Phase 2 Dose (RPTD) and schedule under a 21 day continuous dosing.
Extension Study: Continued assessment of the safety profile of ABT-263 | 21 day continuous dosing
  Continued assessment of the safety profile of ABT-263.
Extension Study: Continued assessment of the preliminary efficacy signals of ABT-263. | day continuous dosing
  Continued assessment of the preliminary efficacy signals of ABT-263.

SECONDARY OUTCOMES:
Phase 1a or Phase 1b safety assessment | Repeating sequence of 14 days on therapy and 7 days off OR 21 day continuous dosing.
  Assessment of the safety of ABT-263
Phase 1a, Phase 1b, or Phase 2a pharmacokinetic profile evaluation | Repeating sequence of 14 days on therapy and 7 days off OR 21 day continuous dosing.
  Evaluation of pharmacokinetic profile of ABT-263.
Phase 1a effect of food on bioavailability | Repeating sequence of 14 days on therapy and 7 days off.
  Evaluation of the effect of food on bioavailability

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, MD, Study Director — AbbVie
Locations (12):
- United States (11):
  - Site Reference ID/Investigator# 4997, Los Angeles, California
  - Site Reference ID/Investigator# 9104, Los Angeles, California
  - Site Reference ID/Investigator# 2613, Bethesda, Maryland
  - Site Reference ID/Investigator# 40243, Boston, Massachusetts
  - Site Reference ID/Investigator# 4745, Boston, Massachusetts
  - Site Reference ID/Investigator# 2628, Buffalo, New York
  - Site Reference ID/Investigator# 23543, New York, New York
  - Site Reference ID/Investigator# 2627, New York, New York
  - Site Reference ID/Investigator# 2614, New York, New York
  - Site Reference ID/Investigator# 5383, New York, New York
  - Site Reference ID/Investigator# 12306, Rochester, New York
- Site Reference ID/Investigator# 8941, Edmonton, Canada

REFERENCES:
- [Background] Wilson WH, O'Connor OA, Czuczman MS, LaCasce AS, Gerecitano JF, Leonard JP, Tulpule A, Dunleavy K, Xiong H, Chiu YL, Cui Y, Busman T, Elmore SW, Rosenberg SH, Krivoshik AP, Enschede SH, Humerickhouse RA. Navitoclax, a targeted high-affinity inhibitor of BCL-2, in lymphoid malignancies: a phase 1 dose-escalation study of safety, pharmacokinetics, pharmacodynamics, and antitumour activity. Lancet Oncol. 2010 Dec;11(12):1149-59. doi: 10.1016/S1470-2045(10)70261-8. Epub 2010 Nov 18. PMID 21094089
- [Derived] de Vos S, Leonard JP, Friedberg JW, Zain J, Dunleavy K, Humerickhouse R, Hayslip J, Pesko J, Wilson WH. Safety and efficacy of navitoclax, a BCL-2 and BCL-XL inhibitor, in patients with relapsed or refractory lymphoid malignancies: results from a phase 2a study. Leuk Lymphoma. 2021 Apr;62(4):810-818. doi: 10.1080/10428194.2020.1845332. Epub 2020 Nov 25. PMID 33236943